CLINICAL TRIAL: NCT04572503
Title: Barbed Suture Modified Anterior Palatoplasty In Management of Mild and Moderate Obstructive Sleep Apnea Syndrome
Brief Title: Modified Anterior Palatoplasty In Obstructive Sleep Apnea Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Abdelrahman Ahmed Abdelalim, MD Lecturer, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS 19-2-2020
Record Dates: First submitted 2020-09-26; First posted 2020-10-01 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Barbed suture; Anterior palatoplasty
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified Anterior Palatoplasty (Experimental): Barbed Suture Modified Anterior Palatoplasty In Management of Mild and Moderate Obstructive Sleep Apnea Syndromea using single resorbable polydioxanone barbed bidirectional size 0 monofilament suture
  Interventions: Procedure: Barbed Suture Modified Anterior Palatoplasty

INTERVENTIONS:
Procedure: Barbed Suture Modified Anterior Palatoplasty — Barbed Suture Modified Anterior Palatoplasty using single resorbable polydioxanone barbed bidirectional size 0 monofilament suture

SUMMARY:
The aim of this study is to evaluate the effectiveness of barbed suture modification of anterior palatoplasty in the treatment of patients with retropalatal mild to moderate obstructive sleep apnea syndrome (OSAS).

DETAILED DESCRIPTION:
A prospective analytic study will be conducted on a total number of 20 patients presented with mild to moderate obstructive sleep apnea for whom Barbed suture modified anterior palatoplasty will be performed.

Surgical Steps

* Procedure will be performed under general anesthesia
* Bilateral tonsillectomy will be performed.
* Then, the inferior portion between upper 2/3 and inferior 1/3 of palatopharyngeus muscle will be partially released
* Then, a rectangular shaped strip of mucosa and the underlying submucosa will be removed at the center of the soft palate consisting of 0.5-0.7 mm in length and with width corresponding to the tonsillar fossae distance.
* Then,the stripped area will be sutured by single resorbable polydioxanone barbed bidirectional size 0 monofilament suture by introducing one needle at the center point of the wound then will be passed laterally within the palate, turning around pterygomandibular raphe till it comes out at the most superior part of the raphe at one side the thread will be pulled until it hangs at the central transition zone which is a free zone present between the two directions of the thread.
* Then, again the needle will be passed back through the tonsillectomy bed and then this suture will be suspended around the raphe again; a gentle traction is then applied on the thread only and no knots are taken.T
* The opposite side will be done by the same way.
* Finally, each thread will be come out at the raphe of the same side, for locking of the stitches and looseness prevention; a superficial stitch in the opposite direction is taken, and then the thread is cut while bushing the tissue downward for more traction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate obstructive sleep apnea syndrome.
* Patients diagnosed with mild (AHI 5 to15) and moderate (AHI 16 to 30) OSAS with only retropalatal collapses
* Patients who are noncompliant with Continuous positive airway pressure (CPAP).

Exclusion Criteria:

* Patients diagnosed with sever OSAS (AHI more than 30)
* The main site of obstruction at retrolingual level or multilevel obstruction.
* Contraindication of surgery (e.g. cardiovascular problems and bleeding tendency).
* Patients with significant craniofacial anomalies affecting airway.
* Patients with BMI>40 kg/m2.
* Patients unfit for general anesthesia.
* History of previous velopharyngeal or lingual surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Apnea Hypopnea index | 6 months
  one-night polysomnographic study at sleep lab. The apnea-hypopnea index denotes the total numbers of apnea plus hypopnea events divided by total sleep time in hours (0-5/ hr sleep = mild, 6-15/hr sleep = moderate, more than 15/hr sleep = severe)

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman A Abdelalim, MD, Principal Investigator — Benha University; Mohamed A Elsayed, MD, Study Chair — Benha University; Hesham A Abdelsamea, MD, Study Chair — Benha University; Ahmed Y Abdelsalam, Resident, Study Chair — Al-Agouza specialized hospital
Locations (1):
- Benha University Hospital, Faculty of Medicine, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pianta L, Bertazzoni G, Morello R, Perotti P, Nicolai P. Barbed expansion sphincter pharyngoplasty for the treatment of oropharyngeal collapse in obstructive sleep apnoea syndrome: A retrospective study on 17 patients. Clin Otolaryngol. 2018 Apr;43(2):696-700. doi: 10.1111/coa.13008. Epub 2017 Nov 6. No abstract available. PMID 29045003
- [Background] Salamanca F, Costantini F, Mantovani M, Bianchi A, Amaina T, Colombo E, Zibordi F. Barbed anterior pharyngoplasty: an evolution of anterior palatoplasty. Acta Otorhinolaryngol Ital. 2014 Dec;34(6):434-8. PMID 25762837